CLINICAL TRIAL: NCT02495753
Title: Vaginal Cleansing Before Cesarean Delivery to Reduce Infection: A Randomized Trial
Brief Title: Vaginal Cleansing Before Cesarean Delivery to Reduce Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201505127
Record Dates: First submitted 2015-06-28; First posted 2015-07-13 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Complications; Cesarean Section
Keywords: cesarean section; wound infection; vaginal cleansing; endometritis
MeSH Terms: conditions — Wound Infection; Endometritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abdominal and Vaginal Cleansing (Experimental): In the treatment arm, the vagina will be cleansed prior to usual abdominal cleansing before cesarean section.
  Interventions: Procedure: Vaginal Cleansing; Procedure: Abdominal Cleansing
- Abdominal Cleansing Alone (Active Comparator): In the control arm, abdominal cleansing will be performed per routine with no vaginal cleansing.
  Interventions: Procedure: Abdominal Cleansing

INTERVENTIONS:
Procedure: Vaginal Cleansing — The vagina will be prepped in two passes with sponge sticks soaked in 1% povidone-iodine solution from a prepackaged sterile pouch.
  Arms: Abdominal and Vaginal Cleansing
Procedure: Abdominal Cleansing — The abdomen will be cleansed using chlorhexidine or betadine according to surgeon's preference prior to cesarean.

SUMMARY:
The purpose of this study is to test the hypothesis that vaginal cleansing with povidone-iodine solution immediately prior to cesarean delivery reduces postcesarean infectious morbidity.

DETAILED DESCRIPTION:
Cesarean delivery is the most common surgical procedure performed on women in the US; nearly 1.3 million are performed each year. Postoperative infectious morbidity is the most common complication of cesarean delivery. Post-cesarean infectious morbidity is often the result of indigenous vaginal flora that ascend into the uterus at the time of surgery. Thus, reducing vaginal microbial load may reduce post-cesarean infection. However, results from studies assessing the role of vaginal cleansing prior to cesarean have been mixed.

The investigators will perform a randomized controlled clinical trial to test the hypothesis that vaginal cleansing with povidone-iodine solution immediately prior to cesarean delivery reduces postcesarean infectious morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing cesarean delivery after labor at Barnes-Jewish Hospital.

Exclusion Criteria:

* Inability to obtain consent
* known or suspected allergy to iodine or shellfish
* women with active herpes simplex virus infection

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2015-08; Primary Completion 2021-01 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Composite Postoperative Infectious Morbidity | 30 days postoperatively
  Maternal fever, endometritis, intrabdominal infection or abscess, wound complication within 30 days of delivery or wound infection.

SECONDARY OUTCOMES:
Adverse Reaction to Vaginal Cleansing | 30 days postoperatively
  Hypersensitivity Reaction or more severe allergic reaction
Length of Hospital Stay | 30 days postoperatively
  Days in hospital
Number of readmissions to hospital for infectious morbidity. | 30 days postoperatively
  Number of times patient is readdmitted for any infectious morbidity.
Treatment for neonatal Sepsis | 30 days postoperatively
  Any antibioitics given for neonate with suspected sepsis.
Number of outpatient visits for infectious morbidiy. | 30 days postoperatively.
  Number of outpatient or emergency room visits related to infectious morbidity.

OTHER OUTCOMES:
Prespecified Stratified Analysis for Subgroups | 30 days postoperatively
  Planned secondary analysis will be aimed at obtaining adjusted assessments of treatment effectiveness with interaction tests used to determine if the effectiveness of vaginal cleansing differs across subgroups. Subgroups include BMI categories, rupture status, chorioamnionitis, stage of labor, cervical dilation >6 cm, gestational age, use of monitors, time in labor, duration of rupture, presence of GBS, labor status, and use of ripening agents.
Prespecified Stratified Analysis for Subgroups | 30 days postoperatively
  Planned secondary analysis will be performed in order to obtain adjusted assessment of treatment effectiveness in subgroups stratified based on the following: administration of azithromycin and time of enrolment date in relation to hospital protocol adjustments for Covid19 screening.

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] Temming LA, Frolova AI, Raghuraman N, Tuuli MG, Cahill AG. Vaginal cleansing before unscheduled cesarean delivery to reduce infection: a randomized clinical trial. Am J Obstet Gynecol. 2023 Jun;228(6):739.e1-739.e14. doi: 10.1016/j.ajog.2022.11.1300. Epub 2022 Nov 30. PMID 36462539
- [Derived] Haas DM, Morgan S, Contreras K, Kimball S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2020 Apr 26;4(4):CD007892. doi: 10.1002/14651858.CD007892.pub7. PMID 32335895